CLINICAL TRIAL: NCT07056140
Title: Effectiveness of Simulation-Based Training for Epidural Analgesia Placement in Obstetric Settings: A Prospective, Randomized, Monocentric Study
Brief Title: Simulation-Based Training for Epidural Analgesia Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 546n/25
Record Dates: First submitted 2025-06-20; First posted 2025-07-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Epidural Analgesia; Medical Education; Obstetric Anesthesia
Keywords: Epidural analgesia; Obstetric anesthesia; Epidural catheter placement; Simulation training; Medical education; Obstetric simulation; Anesthesia training; Technical skills

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: a standard training group or an enhanced simulation-based training group for epidural placement. Each participant will receive only one type of intervention, with no crossover between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Simulator Training Group (Experimental): Participants receive training using the epidural simulator before starting their residency period and actually performing procedures on patients.
  Interventions: Procedure: Epidural Simulation Training; Procedure: Standard Clinical Training
- Traditional Training Group (Active Comparator): Participants receive standard theorical clinical training without the use of the epidural simulator before their residency period in the obstetric unit
  Interventions: Procedure: Standard Clinical Training

INTERVENTIONS:
Procedure: Epidural Simulation Training — The group will have access to a epidural simulator and would have possibility to freely experiment and improve their skill on the phantom before their residency period in the obstetric unit
  Arms: Epidural Simulator Training Group
Procedure: Standard Clinical Training — Participants will receive a standard clinical training based on frontal lessons regarding indications , controindications to epidural analgesia and the technique will be explained also with the use of video material

SUMMARY:
Epidural analgesia is the gold standard for labor pain management, widely recommended by the WHO and included in Italy's essential levels of care (LEA) since 2017. Despite its clinical benefits and high maternal satisfaction, the procedure remains technically challenging, particularly for anesthesia residents. In our institution, around 40% of laboring women request epidural analgesia.

Successful epidural placement requires mastering a complex skillset. Recent studies highlight that simulation-based training significantly enhances learning for novice practitioners. This single-center, prospective, randomized controlled trial aims to evaluate whether a pre-rotation simulator-based training improves the success rate of epidural catheter placement among anesthesia residents.

Participants will be randomly assigned to either the intervention group (simulation training plus anatomy lecture) or the control group (standard in vivo training only). The primary outcome is the number of successful catheter placements (defined as completed procedure without tutor intervention). Secondary outcomes include procedure time, complication rates, and satisfaction scores from the residents. The study will involve anesthesia residents in their 4th or 5th year rotating in the labor ward of the Azienda Ospedaliera di Padova. A sample size of 86 participants (43 per group) is required, and data collection will occur over three years.

DETAILED DESCRIPTION:
Epidural analgesia remains the most effective method to relieve pain during labor. It acts on both visceral and somatic pain pathways and is particularly recommended in various maternal and fetal indications, such as twin pregnancies, induced labor, and high-risk maternal conditions (e.g., obesity, preeclampsia, diabetes). Despite its widespread use, epidural placement is technically demanding, especially in laboring women who are in pain, exhausted, and often overweight.

This complexity is further compounded by the fact that fewer open surgeries are being performed in training settings, which limits residents' opportunities to practice epidural catheter placement under optimal conditions. Hence, the use of simulation-based training has become increasingly important.

The aim of this study is to assess whether prior training with high-fidelity epidural simulators improves the technical success of novice anesthesia residents. Simulation sessions will utilize models already available at the teaching center (Kyoto Kagaku Lumbar Puncture and Epidural Anesthesia Simulators).

This open-label, randomized, single-center interventional study will recruit anesthesia residents with less than 20 previous epidural placements. Residents will be allocated into two groups (simulation vs. control) and further stratified by experience level (novice <20 vs. intermediate >20 prior procedures). Those in the simulation group will receive a frontal anatomy lecture and a 3-hour practical session on simulators before their labor ward rotation.

All procedures will be performed under supervision, and outcome assessors will complete structured CRFs for each attempt. Data will be pseudonymized and stored securely. Analyses will include both parametric and non-parametric tests, with a significance level of p < 0.05. The trial complies with GCP standards and ethical guidelines, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Residents in Anesthesia
* Informed Consent

Exclusion Criteria:

* An experience of 20 or more epidural catheter positioning
* Experience with epidural simulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Epidural Catheter Placement | Immediately following the procedure, up to 45 minutes after the enorllment.
  Defined as successful placement of the epidural catheter in the correct anatomical space as determined by supervising anesthesiologist.

SECONDARY OUTCOMES:
Number of Attempts Required for Successful Placement of the Epidural Cathter | During the procedure, from the enrollment up to 45 minutes after the enorllment
  Total number of needle insertions until successful catheter placement is achieved.
Incidence of Accidental Dural Puncture (Complication) | During the procedure from the enrollment up to 45 minutes after the enorllment
  Number of procedures resulting in unintentional puncture of the dura mater.
Incidence of Bloody Tap (Complication) | During the procedure, from the enrollment up to 45 minutes after the enorllment
  Occurrence of blood in the epidural needle or catheter upon insertion.
Incidence of Supervisor intervention | During the procedure, from the enrollment up to 45 minutes after the enorllment
  The procedure required the attending anesthesiologist intervention to be completed
Success Rate of Epidural Catheter Positioning During the Day Shift | During the procedure, from the enrollment up to 45 minutes after the enorllment
  Defined as successful placement of epidural catheters positioned from 08:00 AM to 08:00 PM in the correct anatomical space as determined by supervising anesthesiologist
Success Rate of Epidural Catheter Positioning During the Night Shift | During the procedure, from the enrollment up to 45 minutes after the enorllment
  Defined as successful placement of epidural catheters positioned from 08:00 PM to 08:00 AM in the correct anatomical space as determined by supervising anesthesiologist
Time to Complete the Epidural Catheter Positioning | From the start to the end of the procedure, from the enrollment up to 45 minutes after the enrollment
  Time to complete the epidural catheter positioning from the skin disinfection to the needle removal

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro De Cassai, Principal Investigator — University of Padova
Locations (1):
- University Hospital of Padua, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided